CLINICAL TRIAL: NCT05160649
Title: Effect of Time of COVID 19 Infection on Fetomaternal Outcome, and Immunological Changes During the Disease Course
Brief Title: Effect of Covid 19 Infection on Fetomaternal Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, lecturer of obstetrics and gynecology Faculty of medicine, Fayoum University
Other Study IDs: S 280
Record Dates: First submitted 2021-12-15; First posted 2021-12-16 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; COVID-19 Pneumonia; Fetal Growth Retardation
Keywords: COVID19 Pneumonia; Feto-maternal infection; COVID 19 placental infection; Maternal mortality; Intrauterine fetal death
MeSH Terms: conditions — COVID-19; Fetal Growth Retardation; Maternal Death; Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The novel coronavirus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was discovered for the first time in December 2019 in Wuhan (China) and the disease it causes is called coronavirus disease 2019 (COVID-19). Now, this pandemic is rapidly spreading all over the world.

Pregnant have higher rates of COVID-19, associated with hospitalizations, and severe in-hospital outcomes. Immune responses may have a potential role in the diagnosis, treatment, and prognosis of patients with COVID-19. So we need of identifying biomarkers for disease severity and progression.

DETAILED DESCRIPTION:
It is important to define whether a novel virus is transmissible from a mother to her infant, vertical infection, and there are three possible mechanisms for vertical infection - intrauterine infection (including transplacental and ascending infections), intrapartum transmission (during delivery), and postpartum infection. These mechanisms have important implications that can influence obstetrical management decisions, best practice delivery options, and neonatal care (3).

Aim of work To detect the effect of time of infection by COVID 19 on the fetomaternal outcome including vertical transmission, and the immunological and genetic changes during the disease course.

Patients and Methods:

* All pregnant women eligible for the study will undergo detailed medical history.
* Each patient will have the following data: • Patient name. • Age. • Past medical and surgical history. • Menstrual history and contraceptive history: especially emphasis on Last Menstrual Period to determine the exact gestational age.
* Clinical examination of the patients: - General examination of vital data (blood pressure, pulse, temperature, respiratory rate). CBC, PT, PTT, RBS, ALT, AST, serum creatinine), and ultrasound will be done.
* Abdominal examination: to detect any abnormality as intrauterine growth restriction, with serial ultrasound estimation.

ELIGIBILITY:
Inclusion Criteria: Pregnant pt with covid 19 infection (at any gestational age) diagnosis of infection based on any one of the following criteria:

1. Positive RT-PCR nasopharyngeal swab is taken (even if the result became available after labor);
2. Positive rapid antigen test performed before labor
3. Chest computed tomography (CT) scan performed before labor showing changes consistent with pneumonitis secondary to SARS-CoV-2 infection;
4. Positive pre-labor immunoglobulin G or immunoglobulin M antibody test; or
5. Clinical diagnosis made before labor (in the absence of negative RT-PCR swab results).

Exclusion Criteria:

1. Healthy individuals:
2. Acute or chronic infectious disease,
3. And any medication with known influence on immunological factors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A prospective observational study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
First, second and third trimester fetomaternal complications. | 3 months
  Abdominal examination: to detect any abnormality as intra uterine growth restriction, with serial ultrasound estimation.
fetal distress | 3 months
  Intrapartum fetal heart rate (FHR) to detect viability and any abnormalities. Pregnant women diagnosed to have intrapartum fetal distress (Non reassuring or pathological changes according to NICE guidelines 2017)

SECONDARY OUTCOMES:
fetal outcome | 3 months
  After birth: Apgar score will be used to identify distress newborns that need resuscitation and nicu admissionsigns of fetal pulmonary complication, acute respiratory distress syndrome.
  The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2. A score of 7 to 10 after five minutes is "reassuring." A score of 4 to 6 is "moderately abnormal." A score of 0 to 3 is concerning. It indicates a need for increased intervention, usually in assistance for breathing.
Time of infection and fetal complications | 3 months
  Time from the diagnosis of SARS-CoV-2 infection to day of labour will be collected as a categorical factor and pre-determined to be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Laila E Abdelfattah, Ass. prof, Principal Investigator — Associated professor of obestatrics and gynecology Faculty of medicine Fayoume university; Eman E Mahmoud, lecturer, Principal Investigator — Lecturer of clinical and chemical pathology
Locations (1):
- Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided